CLINICAL TRIAL: NCT07148895
Title: A Prospective, Randomized, Multi-Center Trial Assessing Post-Operative Outcomes Following Pediatric Sistrunk Procedures With or Without Drain Placement
Brief Title: Assessing Post-operative Outcomes After Children's Sistrunk Procedure With or Without a Drain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Boston Children's Hospital (Other); Connecticut Children's Medical Center (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Jennifer Brooks, Assistant Professor - Department of Otolaryngology (SMD), University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00010365
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Thyroglossal Duct Cysts
Keywords: Sistrunk procedure
MeSH Terms: conditions — Thyroglossal Cyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drain (Active Comparator): During surgery, at the completion of the Sistrunk procedure, participants will have a suction drain placed. The drain will be removed later based on standard criteria prior to discharge from the hospital.
  Interventions: Procedure: Post-surgical drain
- No Drain (Active Comparator): At the completion of the Sistrunk procedure, participants will not have a suction drain placed.
  Interventions: Procedure: No post-surgical drain

INTERVENTIONS:
Procedure: Post-surgical drain — During surgery, at the completion of the Sistrunk procedure, participants in the drain cohort will have a suction drain placed, which will be removed based on standard criteria prior to discharge from the hospital. Wound care following drain removal will be standardized, with instructions for patients to allow the area to heal naturally and to follow a regimen of cleaning and applying topical antibiotic ointment for several days.
  Arms: Drain
Procedure: No post-surgical drain — Patients will be recovered in SOC manner from Sistrunk surgery without drain placement
  Arms: No Drain

SUMMARY:
Purpose of the Study:

This study looks at how kids recover after a type of neck surgery called the Sistrunk procedure. Some kids have a small tube (called a drain) placed during surgery, and some do not. The goal is to see if using a drain makes a difference in how well they heal.

Who Is in the Study:

Children who are having surgery to remove a thyroglossal duct cyst-a common lump in the neck that some kids are born with.

Main Questions the Study Wants to Answer:

Does using a drain lower the chance of problems at the surgery site? Does using a drain change how often kids need more treatment or have to go back to the hospital?

What Will Happen:

Kids will have the Sistrunk surgery, with or without a drain. Doctors will watch how they heal and check for any problems, like infections, needing more procedures, or going back to the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 18 and younger
* Diagnosis of a <3cm midline neck mass, tract or sinus as determined by preoperative physical examination and imaging
* Patient scheduled for Sistrunk procedure (excision of TGDC)
* Patient assigned to the drain or no drain groups at the time of surgery.
* Sistrunk procedure performed per best practices and standardized per surgical study protocol.
* Patient admitted for overnight observation.
* Thyroglossal duct cyst confirmed on final pathology.

Exclusion Criteria:

* Patients with confirmed bleeding or immunodeficiency disorders as previously documented in electronic medical record.
* Lesions greater than 3cm on preoperative ultrasound or axial imaging
* Lingually positioned lesions.
* Evidence of overt infection at the time of surgery
* Coexistent lesion excision (e.g., branchial cleft cyst excision, thyroidectomy)
* Entry into oropharynx noted during procedure.
* Revision surgery if prior formal Sistrunk performed.
* Patients in whom the surgeon deems a drain is necessary.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 178 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Hematoma | 30 days post-procedure
  The occurrence of hematoma will be assessed. A hematoma is defined as a localized collection of blood at the surgical site that is clinically significant and requires management beyond observation (e.g., drainage, surgical evacuation). A single value per participant is derived as yes (hematoma present) or no (hematoma absent). A "yes" indicates a hematoma occurred; a "no" indicates no hematoma occurred.
Occurrence of Seroma | 30 days post-procedure
  The occurrence of seroma will be assessed. A seroma is defined as a localized collection of serous fluid at the surgical site that is clinically significant and requires intervention (e.g., aspiration or drainage). A single value per participant is derived as yes (seroma present) or no (seroma absent). A "yes" indicates a seroma occurred; a "no" indicates no seroma occurred.
Occurrence of Surgical Site Infection (SSI) | 30 days post-procedure
  The occurrence of surgical site infection will be assessed. An SSI is defined as an infection at the surgical site requiring treatment (e.g., antibiotics, wound drainage). A single value per participant is derived as yes (infection present) or no (infection absent). A "yes" indicates an infection occurred; a "no" indicates no infection occurred.

SECONDARY OUTCOMES:
Need for Return to Operating Room (OR) or Procedural Intervention | 30 days post-procedure
  The need for any surgical or procedural intervention related to the Sistrunk procedure will be recorded. A single value per participant is derived as the presence (yes) or absence (no) of an intervention. A "yes" indicates the participant required a return to the OR or procedure; a "no" indicates no intervention was required.
Hospital Readmission | 30 days post-procedure
  Any unplanned hospital readmission lasting greater than 23 hours after initial discharge will be recorded. A single value per participant is derived as yes (readmitted) or no (not readmitted). A "yes" indicates a readmission occurred; a "no" indicates no readmission occurred.
Hospital Length of Stay | 30 days post-procedure
  Hospital length of stay will be measured in total number of days admitted for the index hospitalization. A single value per participant is derived by counting the number of calendar days from admission to discharge. Higher numbers indicate longer hospitalization; lower numbers indicate shorter hospitalization.
Need for Antibiotics | 30 days post-procedure
  Any prescription of antibiotics specifically related to wound healing will be recorded. A single value per participant is derived as yes (antibiotics prescribed) or no (not prescribed). A "yes" indicates antibiotics were required; a "no" indicates antibiotics were not required.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Connecticut Children's, Hartford, Connecticut
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Rochester Medical Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Brooks JA, Cunningham MJ, Hughes AL, Kawai K, Dombrowski ND, Adil E. Postoperative Disposition Following Pediatric Sistrunk Procedures: A National Database Query. Laryngoscope. 2021 Jul;131(7):E2352-E2355. doi: 10.1002/lary.29331. Epub 2021 Jan 11. PMID 33427321
- [Background] Qureshi TA, Suhail A, Zaidi SS, Siddiq W. Is There Any Benefit of Drain Placement on Postoperative Complications in Patients Undergoing the Sistrunk Procedure? Int Arch Otorhinolaryngol. 2015 Oct;19(4):331-5. doi: 10.1055/s-0035-1549156. Epub 2015 Mar 27. PMID 26491480
- [Background] Hong P. Is drain placement necessary in pediatric patients who undergo the Sistrunk procedure? Am J Otolaryngol. 2014 Sep-Oct;35(5):628-30. doi: 10.1016/j.amjoto.2014.04.005. Epub 2014 May 4. PMID 24888796
- [Background] Brooks JA, Cunningham MJ, Koempel JA, Kawai K, Huang JK, Weitzman RE, Osterbauer B, Hughes AL. To drain or not to drain following a Sistrunk procedure: A dual institutional experience. Int J Pediatr Otorhinolaryngol. 2019 Dec;127:109645. doi: 10.1016/j.ijporl.2019.109645. Epub 2019 Aug 19. PMID 31494373
- [Background] Athow AC, Fagg NL, Drake DP. Management of thyroglossal cysts in children. Br J Surg. 1989 Aug;76(8):811-4. doi: 10.1002/bjs.1800760815. PMID 2765833